CLINICAL TRIAL: NCT04300361
Title: A Prospective, Multicenter, Observational Study to Identify Novel Deleterious Variants in the DPYD Gene in Patients of Non-Western Descent: The DPYD-NOW Study
Brief Title: Identifying Novel Variants in the DPYD Gene in Patients of Non-Western Descent
Acronym: DPYD-NOW
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: The Netherlands Cancer Institute (Other); Erasmus Medical Center (Other); Haga Hospital (Other); Medical Center Haaglanden (Other)
Responsible Party: Principal Investigator, HansGelderblom, Prof. dr., Leiden University Medical Center
Other Study IDs: DPNOW
Record Dates: First submitted 2020-02-24; First posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Neoplasms
Keywords: Fluoropyrimidines; DPYD; Genotyping; Capecitabine; 5-Fluorouracil; 5-FU; Non-Western
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. blood sample (whole blood) of 4 ml (EDTA-tube) for sequencing of the DPYD gene
  2. blood samples (whole blood) of 6 ml (EDTA-tubes) each for determination of the DPD enzyme activity
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Non-Western patients: Patients of non-Western descent with an indication for treatment with fluoropyrimidine-based chemotherapy. A patient is classified as non-Western if a one (1) of the parents or more than two (>2) of the grand parents are of non-Western descent.
  Interventions: Genetic: Sequencing of DPYD gene

INTERVENTIONS:
Genetic: Sequencing of DPYD gene — The DPYD gene of non-Western patients will be sequenced to identify DPYD variants that are possibly associated with an increased risk of developing severe fluoropyrimidine-related toxicity.

SUMMARY:
This is a observational, multicenter study to identify novel variants of the DPYD gene which are possible deleterious in patients of non-Western descent.

DETAILED DESCRIPTION:
Research has shown that DPYD-guided dose-individualization based on 4 DPYD variants (DPYD*2A, c.1236G>A, c.2846A>T and c.1679T>G) can significantly reduce severe fluoropyrimidine-related toxicity. However, these 4 variants are most likely not predictive for toxicity in patients of non-Western descent. In this study the DPYD gene of patients of non-Western descent will be sequenced to identify novel variants that could be associated with a reduced DPD enzyme activity and an increased risk of developing severe fluoropyrimdine-related toxicity. Additionally, the ability to predict if a DPYD variant is possibly deleterious by a recombinant model systen (DPYD-varifier) will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed malignancy for which treatment with a fluoropyrimidine is considered to be in the patient's best interest
* Patients need to be self-declared non-Western
* Age 18 years and older
* Able and willing to give written informed consent
* WHO performance status of 0, 1 or 2
* Life expectancy of at least 12 weeks
* Able and willing to undergo blood sampling for study related analysis
* Adequate baseline patient characteristics (complete blood count, hepatic function which involves serum bilirubin, ASAT, ALAT, and renal function)

Exclusion Criteria:

* Prior treatment with fluoropyrimidines
* Patients with known substance abuse, psychotic disorders, and/or other diseases expected to interfere with study or the patient's safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-western patients with an indication for treatment with fluoropyrimidine-based chemotherapy. A patient is classified as non-Western if 1 of the parents or > 2 of the grandparents are of non-Western descent.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Presence of variants of the DPYD gene that are possibly associated with an increased risk of severe fluoropyrimidine-related toxicity in patients of non-Western descent | Patients will be followed for the first 2 cycles (each cycle is 28 days).

SECONDARY OUTCOMES:
DPD enzyme activity of patients carrying a novel DPYD variant compared to wildtype patients measured in peripheral blood mononuclear cells (PBMCs) | Through study completion, an average of 2 years
Ability of the DPYD-varifier to predict if a novel DPYD variant is deleterious | Through study completion, an average of 2 years
Frequency of DPYD variants per ethnic origin | Through study completion, an average of 2 years
Correlation between genetic variants in genes other than DPYD and fluoropyrimidine-related toxicity | Through study completion, an average of 2 years

IPD SHARING:
Plan to Share IPD: No